CLINICAL TRIAL: NCT02334644
Title: A 12-week Randomized Controlled Trial of Probiotic Treatment (Lactobacillus Helveticus R0052 and Bifidobacterium Longum R0175) vs Placebo in Adult Obsessive Compulsive Disorder
Brief Title: Probiotic Treatment in Adult Obsessive-Compulsive Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: drug expired
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-049
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Treatment; Natural Health Product; Anxiety
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Probiotic Formula (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175)
  Interventions: Dietary Supplement: Probiotic Formula (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175)
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Formula (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) — 2 sachets/day x 12 weeks
  Arms: 1
Dietary Supplement: Placebo — 2 sachets/day x 12 weeks
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of 12-weeks of probiotic treatment in adults with primary Obsessive-Compulsive Disorder and whether this treatment will alter the microbiota composition in these patients.

DETAILED DESCRIPTION:
The study will be a prospective, randomized, double blind placebo-controlled trial. The study population will include males and females, ages 18-65, who fulfill criteria for primary DSM-5 OCD as determined by a structured interview. At screening, patients must have a YBOCS score ≥20 and a MADRS score ≤18.

If deemed eligible, patients will provide a stool sample for microbiome profiling and a blood sample for the inflammatory marker analysis. They will return for their first visit where clinician and self-rated symptom severity scales will be completed and patients will begin their randomly assigned treatment condition. Contents of two sachets (probiotic or placebo) will be consumed daily with or just after breakfast.The participants will attend 3 additional study visits, once every 4 weeks and one phone visit at week 6. During these visits, the same clinician and self-reported questionnaires will be completed. At week 6, patients will be contacted by phone to complete the YBOCS and will also provide a midpoint stool sample. At the final visit (week 12) patients will provide a third stool sample for microbiome profiling and a blood sample for inflammatory marker analysis.

Participants will be assessed using the Mini International Neuropsychiatric Interview (MINI) to determine whether criteria for a primary OCD diagnosis is met alongside any additional comorbid disorders.

Participants will complete a number of clinician and self-rated symptom severity scales as listed below:

1. Yale Brown Obsessive-Compulsive Scale (YBOCS) - Clinician-rated
2. Montgomery Asberg Depression Rating Scale (MADRS) - Clinician-rated
3. Obsessive-Compulsive Inventory - Revised (OCI-R) - Self-rated
4. Depression Anxiety Stress Scale (DASS-21) - Self-rated
5. Dutch Dimensional Obsessive-Compulsive Scale (DDOCS) - Self-rated
6. Sheehan Disability Scale (SDS) - Self- rated
7. Quality of Life and Enjoyment Satisfaction Questionnaire - Short Form (Q-LES-Q-SF), Self-rated

   They will also complete additional questionnaires pertaining to their diet and bowel functioning:
8. Gastrointestinal Symptom Rating Scale (GSRS)
9. Short-form Leeds Dyspepsia Questionnaire (SF-LDQ)
10. Rome III criteria for Irritable Bowel Syndrome
11. Assessment of diet using the EPIC-Norfolk Food Frequency Questionnaire.

Subjects will also be asked to provide background information regarding travel in the past 4 months and current place (and duration) of residence as these factors may potentially affect the microbiome profile.

Patients will be weighed and their height measured to determine body mass index (BMI).

Those who meet study criteria will be provided with a collection kit and instructed on appropriate fecal sample collection. Participants will also be given a lab requisition and instructed to have blood drawn at a local lab. This blood sample will examine serum levels of IL-6, IL-1β, IL-10, IFNγ, TNF- α and CRP. Liquid Chromatography-Mass Spectrometry (LC-MS) will be used for a kynurenine/tryptophan analysis.

Fecal Sample Collection Patients and healthy controls will collect fecal samples at home using our well-established protocol. During the recruitment visit, the subjects will be provided a kit containing a single 50-ml sterile vial with an air-tight sachet, and a cooling pad. The stool sample will be brought to the MacAnxiety Research Centre, where it will be stored in -80ºC freezer until the samples are analyzed. All participants will be asked to freeze their samples and deliver them to the MacAnxiety Research Centre 2 weeks following sampling, or earlier.

The visits will be organized as follows:

1. Baseline Visit (visit 1): once blood and stool samples have been collected the patients will be randomized to probiotic or placebo treatment. At this visit patients will begin their randomly assigned treatment condition to probiotic (Lactobacillus helveticus R0052 and Biﬁdobacterium longum R0175) or placebo. The patients will be provided with 60 sachets (probiotic or placebo) and instructed to consume 2 daily sachets with or just after breakfast. At each of the following visit they will be provided with additional 60 sachets.

   In this visit the clinician will also complete the following scales:

   i. Clinical Global Impression - Improvement (CGI-I) - Clinician-rated ii. Clinical Global Impression - Severity (CGI-S) - Clinician-rated iii. Y-BOCS iv. MADRS

   Participants will complete the following scales:
   * Obsessive-Compulsive Inventory - Revised (OCI-R)
   * Depression Anxiety Stress Scale (DASS-21)
   * Dutch Dimensional Obsessive-Compulsive Scale (DDOCS)
   * Sheehan Disability Scale (SDS)
   * Q-LES-Q - short form
2. During the 12 week period of probiotic treatment, subjects will attend 3 additional visits, once every 4 weeks. During each visit (visits 2-4) participants will be assessed by the study physician.

   In each visit the clinician will also complete the following scales:

   i. Clinical Global Impression - Improvement (CGI-I) - Clinician-rated ii. Clinical Global Impression - Severity (CGI-S) - Clinician-rated iii. Y-BOCS iv. MADRS

   Participants will complete the following scales:
   * Obsessive-Compulsive Inventory - Revised (OCI-R)
   * Depression Anxiety Stress Scale (DASS-21)
   * Dutch Dimensional Obsessive-Compulsive Scale (DDOCS)
   * Sheehan Disability Scale (SDS)
   * Q-LES-Q - short form
3. At week 6, patients will provide a midpoint stool sample as per the sample collection protocol outlined above. A member from the research team will also contact the patient via telephone to complete the YBOCS.
4. Visit 4 (week 12): Participants will undergo usual assessment, treatment response will also be determined at this visit (CGI-I score ≤ 2 as well as a 30% drop in YBOCS score). Participants will also complete the Quality of Life and Enjoyment Satisfaction Questionnaire. Patient diet will be assessed using the EPIC-Norfolk Food Frequency Questionnaire. At visit 3, participants will be provided with a collection kit and instructed on appropriate fecal sample collection (as outlined above). The sample should be collected on the prior day to visit 4. Blood samples will be drawn again be drawn at a local lab to examine levels of IL-6, IL-1β, IL-10, IFNγ, TNF- α and CRP. Liquid Chromatography-Mass Spectrometry (LC-MS) will again be used for a kynurenine/tryptophan analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a principal diagnosis of OCD (DSM 5) according to the MINI with a Y-BOCS score of ≥20
2. The ability to comprehend and satisfactorily comply with protocol requirements
3. Written informed consent given prior to beginning of the study.
4. Current use of any psychotropic agent is permitted given that that individual has been on a stable dose for at least 8 weeks.

Exclusion Criteria:

1. Participants with current Major Depressive Disorder.
2. A MADRS score ≥ 18. Patients with significant suicidal ideation (MADRS item 10 ≥ 3) or who have enacted suicidal behaviors within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
3. Individuals with current autoimmune disorders (rheumatoid arthiritis, systemic lupus erythematosus, multiple sclerosis, etc.), inflammatory bowel disease, diabetes.
4. Current use of herbal psychoactive treatments i.e. St. John's Wort, Kava Kava, Chamomile Extract, Valeria. Past use is permitted if treatment ended 3 months prior to entering the study and stool sampling.
5. Participants receiving current psychotherapy, including cognitive behavioural therapy for an anxiety or mood disorder. Past psychotherapy is permitted if treatment ended 3 months prior to entering the study and stool sampling.
6. Patients who currently fulfill criteria for a lifetime history of bipolar disorder, history of drug abuse, a history of schizophrenia or other psychotic disorders, delirium, dementia and amnesic and other cognitive disorders, or are in a current agitated state.
7. Patients meeting criteria for current substance use disorder.
8. Antibiotic or probiotic use within 8 weeks of entering the study and stool sampling.
9. Reports frequent consumption of foods rich in/enriched with probiotics (yogurt etc).
10. Individuals with immune-compromised conditions (i.e. AIDS, lymphoma) or those undergoing long-term corticosteroid treatment.
11. Individuals with a soy or lactose allergy.
12. Female participants must not be breastfeeding, pregnant or seeking to get pregnant during the course of this study.
13. History of allergic response to probiotics or any other related drugs.
14. Currently physically unwell including experiencing nausea, fever, vomiting, abdominal pain, bloody diarrhea.
15. Individuals with prosthetic heart valves, or a history of valvular heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive-Compulsive Scale [YBOCS] | 12 weeks
Clinical Global Impression - Improvement ≤ 2 [CGI-I] | 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline on the following scales: Quality of Life and Employment Satisfaction Questionnaire | 12 weeks
Sheehan Disability Scale | 12 weeks
Montgomery-Asberg Depression Rating Scale (MADRS) | 12 weeks
Obsessive-Compulsive Inventory - Revised | 12 weeks
Depression Anxiety Stress Scale | 12 weeks
Dutch Dimensional Obsessive-Compulsive Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- MacAnxiety Research Centre, Hamilton, Ontario, Canada